CLINICAL TRIAL: NCT05680415
Title: Phase IV Clinical Trial of the Safety, Efficacy, and Immunogenicity of Mycobacterium Vaccae for Injection (Mica) in People Over 15 Years of Age With Latent Mycobacterium Tuberculosis Infection
Brief Title: Clinical Trial of Mica
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LKM-2022-BWK01
Record Dates: First submitted 2022-11-27; First posted 2023-01-11 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Latent Tuberculosis Infection
MeSH Terms: conditions — Latent Tuberculosis | interventions — Injections

STUDY DESIGN:
Intervention Model Description: The experimental group and the blank control group were randomly assigned in a ratio of 1:1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Mycobacterium vaccae for injection (Mica) :
  Dosage form: injection. Main ingredients and contents:Mycobacterium protein 22.50μg/ bottle. Open the aluminum-plastic combination cap of the Xilin bottle, dilute it with 1.0ml sterilized water for injection, shake well, extract the liquid, and inject it deep into the buttocks muscle. Six times every two weeks.
  Interventions: Biological: Mycobacterium Vaccae for Injection
- Blank Group (No Intervention): Non-injection drug.

INTERVENTIONS:
Biological: Mycobacterium Vaccae for Injection — The experimental group was alternately injected with 1 dose of microcard every two weeks (0-2-4-6-8-10 weeks) in the left and right hip muscle deep, and a total of 6 doses were injected.
  Arms: Treatment Group

SUMMARY:
This study used a randomized, open, blank control design. A total of 6800 patients over 15 years old with latent mycobacterium tuberculosis infection who met the inclusion criteria but did not meet the exclusion criteria were randomly assigned to the experimental group and the blank control group in a 1:1 ratio, with 3400 patients in each group. The experimental group was alternately injected with 1 dose of microcard every two weeks (0-2-4-6-8-10 weeks) in the left and right hip muscle deep, with a total of 6 doses. The blank control group was not injected with drugs.

DETAILED DESCRIPTION:
1. Effectiveness evaluation

   Chest imaging examinations were performed at 6, 12, 18 and 24 months after full injection. The blank control group underwent chest imaging examination at 6, 12, 18 and 24 months after 10 weeks. The confirmed and clinically diagnosed cases of tuberculosis in the experimental group were collected from the first dose to 24 months after full injection and the blank control group from 24 months +10 weeks after enrollment. Follow-up is completed if 8 confirmed cases have been collected after 24 months. If no cases are collected within 24 months, follow-up is required until 8 confirmed cases are collected, and follow-up after 24 months only requires chest imaging every 6 months.
2. Safety evaluation

   In the experimental group, AE was collected 30 minutes after each dose, AE was collected from the first dose to 30 days after the full dose, and SAE and AESI (including immune system related diseases such as thyroid/parathyroid disease) from the first dose to 6 months after the full dose. All pregnancy events from the first dose to 30 days after the full dose were collected.

   In the control group, only all AESI (including immune system related diseases such as thyroid/parathyroid diseases) were collected up to 10 weeks and 6 months of enrollment.

   The test group underwent thyroid palpation examination before injection and 6 months after injection. The blank control group underwent thyroid palpation examination on the day of enrollment, 10 weeks and 6 months after enrollment. Cervical ultrasound examination and five tests of thyroid function were added if there were abnormal thyroid palpation in the experimental group at 6 months after full injection and the blank control group at 10 weeks +6 months.
3. Immunogenicity evaluation

Blood samples of the first 100 subjects in the experimental group and the control group were collected for immunogenicity evaluation, which included cellular immunity and humoral immunity. The first 25 subjects in each group were tested for the absolute number of total white blood cells and specific T cells per unit volume of blood. Blood collection time points: 1 month and 12 months before the first dose of the experimental group was injected; The blank control group was the day of enrollment, 1 month +10 weeks and 12 months +10 weeks after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15 and above (≥15 years old), gender unlimited;
2. I (and my guardian) agree to participate in this study and sign the informed consent, willing and able to comply with the requirements of the clinical study protocol;
3. Patients with normal body temperature (axillary temperature < 37.3℃);
4. The mean diameter of the skin test of recombinant mycobacterium tuberculosis fusion protein (EC) is not less than 5mm, or there are blisters, necrosis, lymphangiitis.

Exclusion Criteria:

1. Patients with a history of severe drug allergy, vaccine allergy, allergic constitution or known allergy to experimental drugs;
2. Patients currently suffering from tuberculosis;
3. Acute fever diseases, infectious diseases (including but not limited to measles, whooping cough, influenza, pneumonia, etc.), diabetes mellitus with complications, acute or progressive liver or kidney disease, acute conjunctivitis of the eye, acute otitis media, severe heart disease, severe hypertension, myocardial damage, significant vascular sclerosis, patients with endocarditis, patients with malignant tumors, etc.;
4. Patients with extreme weakness and severe anemia;
5. Patients with a history of convulsions, epilepsy, encephalopathy, and neurological symptoms or signs upon examination;
6. Chest imaging examination showed active tuberculosis;
7. Patients with abnormal thyroid palpation or a history of thyroid/parathyroid disease;
8. The interval between other subunit vaccines and inactivated vaccines was less than 7 days, and the interval between attenuated live vaccines was less than 14 days before enrollment;
9. Women who are pregnant or breastfeeding, who test positive for pregnancy, or who cannot guarantee contraception during the study period of this clinical trial;
10. Any circumstances which the investigator considers likely to influence the evaluation of the test.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6800 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
End point of efficacy | through study completion, an average of 2 year
  Subjects were monitored for confirmed TB cases from enrollment to 24 months after the completion of the injection.

SECONDARY OUTCOMES:
End point of safety | 30 minutes and 30 days after each dose
  The number of cases of all adverse events occurring within 30 minutes and 30 days after each dose.
End point of safety | 6 months after the first dose to the full dose
  Incidence of SAE and AESI within 6 months after the first dose to the full dose
End point of immunogenicity | Treatment group: 1 month and 12 months before drug injection, after full injection; Blank control group: the day after enrollment, 1 month +10 weeks after enrollment, 12 months +10 weeks.
  Humoral Immunity:Changes in the amount of total IgG antibody and IgG subclasses (IgG1 and IgG2).
End point of immunogenicity | Treatment group: 1 month and 12 months before drug injection, after full injection; Blank control group: the day after enrollment, 1 month +10 weeks after enrollment, 12 months +10 weeks.
  Cellular immunity: PBMCs antigen-specific IFN-γ level changes;
End point of immunogenicity | Treatment group: 1 month and 12 months before drug injection, after full injection; Blank control group: the day after enrollment, 1 month +10 weeks after enrollment, 12 months +10 weeks.
  Cellular immunity: Antigen-specific T cells: the ratio of CD4+ T cells, CD8+ T cells and CD3+ T cells changed;
End point of immunogenicity | Treatment group: 1 month and 12 months before drug injection, after full injection; Blank control group: the day after enrollment, 1 month +10 weeks after enrollment, 12 months +10 weeks.
  Cellular immunity: Changes in the absolute number of total white blood cells and specific T cells per unit volume of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Mo, Master, Principal Investigator — Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Liujiang district Prevention and Control center, Liuchow, Guangxi
  - Liuzhou Center for Disease Control and Prevention, Liuchow, Guangxi